CLINICAL TRIAL: NCT04347681
Title: A National Collaborative Multicenter Phase II Study for Potential Efficacy of Convalescent Plasma to Treat Severe COVID-19 and Patients at High Risk of Developing Severe COVID-19
Brief Title: Potential Efficacy of Convalescent Plasma to Treat Severe COVID-19 and Patients at High Risk of Developing Severe COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King Fahad Specialist Hospital Dammam (Other)
Collaborators: King Fahad Medical City (Other Government); King Faisal Specialist Hospital & Research Center (Other); King Abdulaziz Medical City (Other Government); King Fahad University Hospital (Unknown); John Hopkins Aramco Healthcare (Unknown); Taibah University (Other); King Saud University (Other); King Khaled University Hospital (Unknown); King Fahad Military Medical Complex (Unknown); Qatif Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAEM0321
Record Dates: First submitted 2020-04-08; First posted 2020-04-15 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Convalescent Plasma for COVID 19

STUDY DESIGN:
Intervention Model Description: experimental arm receiving convalescent plasma and parallel arm is control.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): We are aiming to include 40 patients (recipients) who have COVID 19 but have not recovered yet as per the inclusion criteria.
  Interventions: Other: convalescent plasma from recovered COVID 19 donor
- control group (No Intervention): Patients who only consent for sharing their clinical and laboratory data will serve as a control group to compare the efficacy of the convulsant plasma. Age and sex matched historical control could be used if need.

INTERVENTIONS:
Other: convalescent plasma from recovered COVID 19 donor — After obtaining informed consent, Eligible Patients who have severe COVID-19 and have not recovered yet will be infused with the donated convalescent plasma (10-15 ml/kg body weight of recipient)19 at least once & if possible, daily, for up to 5 sessions.
  Arms: Treatment Group

SUMMARY:
Coronavirus disease (COVID-19) pandemic has started to affect Saudi Arabia and is expected to cause a lot of morbidities and many patients, especially the elderly, will require intensive care unit (ICU) support to survive as its lethality increases with the increasing age. Development of a vaccine by pharmaceutical companies like Roche and antibody concentrates from convalescent patients' plasma by Takeda will take 10-12 months to complete, and we speculate that it will be overwhelmingly expensive and limited in supply. We are presenting this urgent proposal to use the convalescent plasma to save the lives of severely affected COVID-19 patients. Most of the logistic support is already available in MOH Saudi Arabia, and it will be a cheap and quick technique based on the time-tested principles of passive immunization which is supported by the most recent data from China. We are proposing to test the therapeutic potential of convalescent plasma (from patients who have fully recovered from COVID-19) in treating patients with serious COVID-19 disease or those who are at risk of developing a serious disease based on their comorbidities profile. Convalescent plasma could provide our first-line defense for people with Covid-19, especially those who are older and at a much higher risk for complications. Amid the COVID-19 pandemic, with no available vaccine or proven antiviral drug, antibodies from recovering patients could provide a "stopgap" measure to help in controlling the pandemic effects on health and economy.

We plan to recruit at least 40 consenting donors and patients. Non-consenting patients will serve as controls.

DETAILED DESCRIPTION:
Coronaviruses (CoV) are a large family of RNA viruses that cause illnesses ranging from the common cold to more severe diseases such as Middle East Respiratory Syndrome (MERS-CoV) and Severe Acute Respiratory Syndrome (SARS-CoV).1,2 The new strain of coronavirus identified in December 2019 in Wuhan city, Hubei province of China, was called 2019 novel coronavirus (2019- nCoV) and has been named by the International Committee on Taxonomy of Viruses (ICTV) as Severe Acute Respiratory Syndrome Corona Virus-2 (SARS-CoV-2). The ICTV have determined that SARS-CoV-2 is the same species as SARS-CoV but a different strain. The World Health Organization (WHO) has named the disease associated with SARS-CoV-2 infections as "COVID-19".

Clinical features of SARS-CoV-2 infection typically include respiratory symptoms, fever, cough, shortness of breath and breathing difficulties. In more severe cases, the infection can cause pneumonia, severe acute respiratory distress syndrome (ARDS), kidney failure and even death. It is not easy to differentiate between non-SARS-CoV-2 seasonal influenza and other respiratory viruses including the locally reported MERS-CoV and H1N1 influenza viruses. SARS-CoV-2 has a higher transmission rate (TR) with an approximate fatality rate of 3%. Although most of the younger patients recover after milder disease, but COVID-19 is most aggressive in the elderly population with worst pneumonia and death rates may reach 14.8%.4 Final diagnosis of SARS-CoV-2 infection depends on viral detection (and if possible, exclusion of other viruses e.g. by Respiratory Viral Panel). Laboratory detection of the SARS-CoV2 is based on detection of viral RNA by real-time reverse transcription-polymerase chain reaction (rRT-PCR) with confirmation by nucleic acid sequencing when necessary.1-5 For example, GeneFinder™ COVID-19 Plus RealAmp Kit is the One-Step Reverse Transcription Real-Time PCR Kit designed to detect the Novel Coronavirus (COVID-19) qualitatively through Reverse Transcription reaction and Real-Time Polymerase Chain Reaction. We will use this or equivalent method to confirm the diagnosis and will repeat the rRT-PCR to make sure it has become negative in a recovered patient. As of now, no vaccine or antiviral drug coming soon, antibodies from recovering patients could provide a "stop-gap" measure to help in controlling the pandemic. The concept of using convalescent plasma is not new. It has been tried in limited numbers of patients during more-recent viral crises, including the 2003 SARS (severe acute respiratory syndrome) epidemic, the 2009 "swine flu" epidemic, and the 2012 outbreak of MERS (Middle East respiratory syndrome).6 Convalescent plasma treatment reduced mortality in patients with severe pandemic influenza A (H1N1) 2009 Virus Infection.7 Patients with a resolved viral infection will develop a polyclonal antibody immune response to different viral antigens of 2019-nCoV. Some of these polyclonal antibodies will likely neutralize the virus and prevent new rounds of infection, and the patients with resolved infection should produce 2019-nCoV antibodies in high titer. Patients with resolved cases of 2019-nCoV can simply donate plasma, and then this plasma can be transfused into infected patients.8 Given that plasma donation is well established, and the transfusion of plasma is also routine medical care, this proposal does not need any new science or medical approvals in order to be put into place. Indeed, the same rationale was used in the treatment of several Ebola patients with convalescent serum during the outbreak in 2014-2015.9 Since the emergence of this SARS-CoV-2 infection in Wuhan, China, in December 2019, it has rapidly spread across China and more than 188 other countries and territories. According to the WHO, as of March 27, 2020, there have been 540,832 confirmed cases worldwide and 24,294 deaths. SARS-CoV-2 has structural similarity to SARS-CoV that caused SARS and MERS-CoV.3 In the Kingdom of Saudi Arabia, there are 1012 confirmed cases reported till now, with 3 deaths (on March 26, 2020).

The Saudi government's prompt actions to slow down the spread of SARS-CoV-2 seem to be effective. However, CDC Estimates 40-70% of the US population will be infected with SARS-CoV-2. Even with curtailment measures, judging from past pandemics, approximately 40% of human beings will be exposed to COVID-19 over the next 2-3 years. Most of these infected people will recover and almost all of them will be immune. Vigilance and readiness are needed to teach the masses about preventive measures because older people and those with comorbidities will be the sickest. Contemporaneously, therapeutic measures are highly needed from the medical community to treat COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:s

1. Recipients:

   We will use the confirmed case definition of SARS-CoV-2 infection (COVID-19) with POSITIVE rRT PCR test for SARS-CoV-2 "using one of the SFDA approved kit used in KSA" as per current MOH / SCDPC (Waqayah) guidelines (derived from WHO and CDC ).
   1. 18 or older
   2. Patient with COVID 19 confirmed as per case definition of CDC or MOH/Waqayah
   3. Must have been requiring ICU care or severe or immediately life-threatening care:

   i. Patient requiring ICU admission. ii. Severe disease is defined as:
   1. Dyspnea
   2. Respiratory frequency ≥ 30/min
   3. Blood oxygen saturation ≤ 93%
   4. Partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300, and/or Lung infiltrates > 50% within 24 to 48 hours iii. Life-threatening disease is defined as:

   <!-- -->

   1. Respiratory failure
   2. Septic shock, and/or
   3. Multiple organ dysfunction or failure
2. Donors:

   1. 18 or older
   2. Recovery from Prior confirmed COVID-19 diagnosis through NEGATIVE rRT PCR test for SARS-CoV-2 from blood or nasopharyngeal swab - FDA IND guidance or the MOH updated recovery protocol 15.20.22.23
   3. Complete Clinical Recovery from COVID-19 at least 14 days prior to donation (FDA IND guidance15)
   4. All MOH criteria for a fit donor will be followed prior to donation.
   5. All Transfusion Transmissible Infections (TTI) markers on the donor blood are negative as per current MOH routine donor screening regulations

Exclusion Criteria:

1. Recipients:

   1. Negative or non-conclusive test COVID-19 rRT PCR test for SARS-CoV-2
   2. Mild symptoms
   3. Hospitalization not requiring ICU admission
2. Donors:

   1. Unfit to donate.
   2. Multiparous or pregnant females.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 575 (Actual)
Dates: Start 2020-04-18 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
ICU length of stay | Time from transfer into ICU to time of transfer out from ICU, Up to 12 weeks.
  number of days in ICU
Safety of convalescent plasma & Serious adverse reactions. | time from signing consent to one month after transfusion, Up to 12 weeks.
  reporting adverse events associated with transfusion as per transfusion medicine guidelines.

SECONDARY OUTCOMES:
Number of days on mechanical ventilation | Time from intubation to time of extubation, Up to 12 weeks.
  number of days patient spend on ventilator.
30 days of mortality | 30 days from signing consent Up to 12 weeks.
  the death rate in 30 days after signing consent
Days to clinical recovery . | time from signing consent to recovery,Up to 12 weeks.
  number of days to symptoms resolution and COVID 19 negative PCR ( by NP swap)

CONTACTS AND LOCATIONS:
Overall Officials: Hani Al-Hashmi, MD, Principal Investigator — King Fahad Specialist Hospital
Locations (14):
- Saudi Arabia (14):
  - John Hopkins Aramco Healthcare, Dhahran, Eastern Provence
  - Qatif Central Hospital, Al Qaţīf
  - Dammam Medical Complex, Dammam
  - Imam Abdulrahman Bin Faisal University, Dammam
  - king Fahad specialist hospital, Dammam
  - DHahran Military Medical Complex, Dhahran
  - International Medical Center, Jeddah
  - Madinah General Hospital, Madinah
  - Ohud Hospital, Madinah
  - Taibah University, Madinah
  - King Abdulaziz Medical City, Riyadh
  - King Fahad Medical City, Riyadh
  - King Faisal Specialist Hospital & Research Center, Riyadh
  - King Khalid University Hospital, Riyadh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] AlShehry N, Zaidi SZA, AlAskar A, Al Odayani A, Alotaibi JM, AlSagheir A, Al-Eyadhy A, Balelah S, Salam A, Zaidi ARZ, Alawami D, Alshahrani MS, AlMozain N, Abulhamayel YM, Al Qunfoidi R, Alfaraj M, Qushmaq N, Alansari R, Dayel A, Elgohary G, Al Bahrani A, Nabhan Abdelhameed AA, AlZahrani HA, Alturkistani H, AlShehry N, Albalawi MA, Elalfy I, Alhumaidan H, Al-Hashmi H; KSA COVID-19 Convalescent Plasma Study Group. Safety and Efficacy of Convalescent Plasma for Severe COVID-19: Interim Report of a Multicenter Phase II Study from Saudi Arabia. Saudi J Med Med Sci. 2021 Jan-Apr;9(1):16-23. doi: 10.4103/sjmms.sjmms_731_20. Epub 2020 Dec 26. PMID 33519339
- [Derived] Albalawi M, Zaidi SZA, AlShehry N, AlAskar A, Zaidi ARZ, Abdallah RNM, Salam A, AlSagheir A, AlMozain N, Elgohary G, Batarfi K, Alfaraedi A, Khojah O, Al-Ansari R, Alfaraj M, Dayel A, Al Bahrani A, Abdelhameed AN, Alhumaidan H, Al-Otaibi JM, Radwi G, Raizah A, Shatry H, Alsaleh S, AlZahrani H, Al-Hashmi H. Safety and Efficacy of Convalescent Plasma to Treat Severe COVID-19: Protocol for the Saudi Collaborative Multicenter Phase II Study. JMIR Res Protoc. 2020 Oct 2;9(10):e23543. doi: 10.2196/23543. PMID 32903199